CLINICAL TRIAL: NCT00621374
Title: Pilot Study of CBT and Self-hypnosis Training for Pain in Persons With Multiple Sclerosis
Brief Title: Management of Pain in Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Mark Jensen, Principal Investigator, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 32022-A; NMSS Award# PP1465
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Multiple Sclerosis; Pain
Keywords: Pain Management; Cognitive Behavior Therapy; Hypnosis
MeSH Terms: conditions — Multiple Sclerosis; Pain; Agnosia | interventions — Cognitive Behavioral Therapy; Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Random Order 1 (Experimental): Randomization Order 1= 1)CONT, 2)CBT, 3)HYP, 4) CBT-HYP
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT) +Hypnosis (HYP); Behavioral: Cognitive Behavioral Therapy (CBT); Behavioral: Self-Hypnosis Training (HYP); Behavioral: Education Control (CONT)
- Random Order 2 (Experimental): Randomization order 2= 1)CONT, 2)HYP, 3)CBT, 4) CBT-HYP
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT) +Hypnosis (HYP); Behavioral: Cognitive Behavioral Therapy (CBT); Behavioral: Self-Hypnosis Training (HYP); Behavioral: Education Control (CONT)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) +Hypnosis (HYP) — There is also the possibility that the two treatments together may be even more helpful than either one alone. Because some of the patients in this study will get both CBT and self-hypnosis, we will be able to determine if each one facilitates the efficacy of the other. If the patients treated in this study report benefits, as we expect they will, then this will encourage us to design and complete a larger study to better understand how patients with MS would benefit from these treatments.
Behavioral: Cognitive Behavioral Therapy (CBT) — One treatment module is we will study is called "cognitive restructuring" or "cognitive-behavior therapy" (CBT). In this treatment, people learn to identify negative thoughts that make them feel bad or anxious. Such negative thoughts lead to feelings of frustration and anxiety, and can even increase the experience of pain, because they cause a person to focus more on pain. With CBT, people learn to identify and stop these thoughts, and then replace them with more reassuring ones. When they do this, they feel more relaxed and focus less on their pain. As a result, they often say that they feel much better and are less aware of pain.
Behavioral: Self-Hypnosis Training (HYP) — Self-hypnosis (HYP) is another strategy that people can learn to manage pain. With this treatment, people learn to enter a state of focused attention, and then change how they experience pain. Although we do not yet know how hypnosis works, research has repeatedly shown that the effects are real; when people report decreases in pain with hypnosis, scans and images of the brain's activity show decreases in the parts of the brain that process pain information. With hypnosis, people are not just pretending to feel less pain, they actually do feel less pain.
Behavioral: Education Control (CONT) — The CONT condition for this study will include lectures that are interactive and are compelling and informative enough to be both (1) credible as an attentional control condition and (2) perceived as helpful to subjects. The CONT condition will not, however, include instructions in making specific cognitive or behavioral changes related to pain management. Thus, it could control for non-specific factors related to behavioral treatment, but will not impact the primary outcome measure (pain).

SUMMARY:
The purpose of this study is to see if treatments that include components of self-hypnosis training and cognitive behavioral therapy (CBT) can help decrease pain in people with MS.

DETAILED DESCRIPTION:
This study examined the benefits of two treatments, individually and together, for helping individuals with MS manage their pain. We conducted a time series design in which MS subjects received all four treatment conditions in two orders (randomly assigned): (1) Control (education intervention-CONT),Self-Hypnosis Training (HYP), Cognitive Behavioral Therapy (CBT), HYP-CBT(a combination of HYP and CBT) and (2) CONT, CBT, HYP, HYP-CBT. Subjects attended 16 60-minute treatment sessions conducted by one of the study's psychologists either at the UW,HMC or in the subject's home. Each subject received four treatment sessions of each treatment module listed above. Primary outcome measures were collected via the telephone and mail by research personnel blind to the treatment condition before treatment, immediately after treatment ends and one month after treatment ends. Secondary outcome measures were collected at the same assessment points via pencil and paper interviews completed by subjects.

ELIGIBILITY:
Inclusion Criteria:

* Chronic ongoing pain (i.e., pain at all times) with an average pain intensity of at least 4/10 on 0-10 numeric rating scale
* Pain is either worse or started since the onset of other MS symptoms.
* Pain of at least six months duration.
* Reads, speaks and understands English.
* Definitive diagnosis of multiple sclerosis (MS)
* At least 18 years of age
* Recruited from a recruitment source approved by the IRB

Exclusion Criteria:

* Severe cognitive impairment resulting in the inability to verbally comprehend, learn, and recall new auditory verbal information, as reflected by a TICS score of 20 or less.
* Currently participating in counseling and/or psychotherapy more than once a week.
* Currently taking anti-psychotic medications
* Has been hospitalized for psychiatric reasons in the past six months
* Experiencing current active suicidal ideation.
* Has received treatment or participated in a clinical trial that involved significant elements of either CBT or hypnosis within the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
A composite of average daily pain intensity measured using a 0-10 NRS via four phone interviews performed on different days by research staff. | Before treatment, after each treatment module, and 1-month after the final treatment module.

SECONDARY OUTCOMES:
Sleep quality- Medical Outcomes Sleep Study Measure (Hays et al., 2005) | before treatment, after each treatment module, one month after 4th treatment modules
Depression- (CMDI; Nyenhuis et al., 1998) | before treatment, after each treatment module, one month after 4th treatment modules
Catastrophizing cognitions- (PCS; Sullivan et al. 1995) | before treatment, after each treatment module, one month after 4th treatment modules
Adaptive cognitions (CPAQ; McCracken et al., 2004) | before treatment, after each treatment module, one month after 4th treatment modules
Distinguishing neuropathic vs. non-neuropathic pain (S-LANSS; Bennett et al., 2005) | before treatment, after each treatment module, one month after 4th treatment modules
Pain Interference-(Brief Pain Inventory, Cleeland et al., 1994) | before treatment, after each treatment module, one month after 4th treatment modules
Impact of Fatigue (FIS; Fisk et al. 1993) | before treatment, after each treatment module, one month after 4th treatment modules
Fatigue Severity (FSS; Krupp et al., 1989) | before treatment, after each treatment module, one month after 4th treatment modules
Health Status (SF-36; Ware et al., 1992) | before treatment, after each treatment module, one month after 4th treatment modules

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Jensen, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Jensen MP, Ehde DM, Gertz KJ, Stoelb BL, Dillworth TM, Hirsh AT, Molton IR, Kraft GH. Effects of self-hypnosis training and cognitive restructuring on daily pain intensity and catastrophizing in individuals with multiple sclerosis and chronic pain. Int J Clin Exp Hypn. 2011 Jan;59(1):45-63. doi: 10.1080/00207144.2011.522892. PMID 21104484